CLINICAL TRIAL: NCT01830855
Title: A Phase 3, Randomized, Active-controlled, Observer-blinded Trial To Assess The Lot Consistency, Safety, Tolerability, And Immunogenicity Of A Meningococcal Serogroup B Bivalent Rlp2086 Vaccine In Healthy Subjects Aged >/=10 To <19 Years
Brief Title: A Trial to Assess the Lot Consistency, Safety, Tolerability and Immunogenicity of Bivalent rLP2086 Vaccine When Given to Healthy Subjects Aged ≥10 to <19 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1971009; 6108A1-3001 (Other: Alias Study Number); 2010-023873-20 (EudraCT Number)
Record Dates: First submitted 2013-04-03; First posted 2013-04-12 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Meningococcal Vaccine
MeSH Terms: interventions — factor H-binding protein, Neisseria meningitidis; Hepatitis A Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rLP2086 lot 1 (Experimental)
  Interventions: Biological: rLP2086
- rLP2086 lot 2 (Experimental)
  Interventions: Biological: rLP2086
- rLP2086 lot 3 (Experimental)
  Interventions: Biological: rLP2086
- Control (Active Comparator): Havrix (HAV) and Saline
  Interventions: Biological: Havrix (HAV); Biological: Saline

INTERVENTIONS:
Biological: rLP2086 — 0.5 mL dose, given at 0, 2 and 6 months (lot 1)
  Arms: rLP2086 lot 1
Biological: rLP2086 — 0.5 mL dose, given at 0, 2 and 6 months (lot 2)
  Arms: rLP2086 lot 2
Biological: rLP2086 — 0.5 mL dose, given at 0, 2 and 6 months (lot 3)
  Arms: rLP2086 lot 3
Biological: Havrix (HAV) — 0.5 mL dose or 1.0 mL dose dependent on age given at month 0 and 6.
  Arms: Control
Biological: Saline — 0.5 mL dose of sterile normal saline for injection.
  Arms: Control

SUMMARY:
This study is looking at a new vaccine that might prevent meningococcal disease, and will study whether healthy adolescent subjects receiving different lots of vaccine respond in a similar way. The study will also look at the safety of the new vaccine as well as how it is tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged >=10 and <19 years at the time of enrollment.
2. Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
3. Negative urine pregnancy test for all female subjects.

Exclusion Criteria:

1. Previous vaccination with any meningococcal serogroup B vaccine.
2. Subjects who have received prior HAV vaccination.
3. Subjects who are scheduled to receive 1 or more doses of an HPV vaccine as part of a 3-dose series during the period between Visit 1 and 28 days after the second vaccination.
4. Subjects receiving any allergen immunotherapy with a nonlicensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
5. A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function, those receiving chronic systemic (oral, intravenous, or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects in the United States with terminal complement deficiency are excluded from participation in this study.
6. Significant neurological disorder or history of seizure (excluding simple febrile seizure).
7. Current chronic use of systemic antibiotics.
8. Received any investigational vaccines, drugs, or devices within 28 days before administration of the first study vaccination.
9. Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3596 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (97):
- United States (60):
  - Birmingham Pediatric Associates, PC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Southeastern Pediatrics, Dothan, Alabama
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - California Research Foundation, San Diego, California
  - Colorado Springs Health Partners/Clinical Research Advantage, Inc., Colorado Springs, Colorado
  - Aga Clinical Trials, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Accelovance, Melbourne, Florida
  - North Georgia Clinical Research Center, Dalton, Georgia
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Accelovance, Inc., Mishawaka, Indiana
  - Optimal Research, LLC, Mishawaka, Indiana
  - Nassim, McMonigle, Mescia & Associates, New Albany, Indiana
  - Augusta Family Practice, Augusta, Kansas
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Central Kentucky Research Associates, Inc., Mount Sterling, Kentucky
  - Mt. Sterling Pediatrics, Mount Sterling, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - David B. Ware, MD, Eunice, Louisiana
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - ACC Pediatric Research, Haughton, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - Southwestern Medical Clinic Lakeland HealthCare Affiliate, Niles, Michigan
  - Allina Health Bandana Square Clinic, Saint Paul, Minnesota
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Bellevue Urgent Care, Bellevue, Nebraska
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Meridian Clinical Research, Llc, Omaha, Nebraska
  - Winthrop Division of Pediatric Infectious Diseases, Mineola, New York
  - Winthrop Pediatric Associates, Mineola, New York
  - Winthrop University Pharmacy, Mineola, New York
  - Winthrop-University Hospital - Clinical Trials Center, Mineola, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Asheboro Research Associates, Asheboro, North Carolina
  - Cary Pediatric Center, Cary, North Carolina
  - Capitol Pediatrics & Adolescent Center PLLC, Raleigh, North Carolina
  - Dr. Shelly David Senders, MD Inc. dba Senders Pediatrics, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Ohio Pediatrics, Inc., Dayton, Ohio
  - Liberty Family Practice, Erie, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Uniontown, Pennsylvania
  - PEAK Research, LLC, Upper Saint Clair, Pennsylvania
  - Holston Medical Group - Suite 3B, Kingsport, Tennessee
  - Holston Medical Group Laboratory, Kingsport, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Cumberland Pediatrics Associates, Lebanon, Tennessee
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Pediatric Research of Charlottesville, Charlottesville, Virginia
  - Advanced Pediatrics, Vienna, Virginia
  - The Vancouver Clinic, Vancouver, Washington
- Canada (5):
  - Medicor Research Inc., Greater Sudbury, Ontario
  - Dr. Hartley Garfield Medicine Professional Corporation, Toronto, Ontario
  - Clinique Medicale St-Louis (recherche) Inc., Québec, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Czechia (8):
  - Ordinace praktickeho lekare pro deti a dorost, Brandýs nad Labem-Stará Boleslav
  - Fakultni nemocnice Hradec Kralove, Klinika infekcnich nemoci,Centrum ockovani a cestovni mediciny, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Hradec Králové
  - Ordinace praktickeho lekare pro deti a dorost, Jindřichův Hradec
  - Ordinace praktickeho lekare pro deti a dorost, Odolena Voda
  - MUDr. Elena Adamkova, Pardubice
  - Zdravotnicke stredisko Dubina v.o.s., Pardubice
  - Ordinace praktickeho lekare pro deti a dorost, Prague
- Finland (4):
  - Helsinki East Vaccine Research Clinic, Helsinki
  - Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - Oulu Vaccine Research Clinic, Oulu
  - Vantaa East Vaccine Research Clinic, Vantaa
- Germany (3):
  - Central Laboratory and Vaccination Centre, Stiftung Juliusspital, Würzburg, Bavaria
  - Kinderarztpraxis Dr. Thomas Adelt, Bramsche
  - Gemeinschaftspraxis für Kinder- und Jugendmedizin Dres. Behre, Burgert, Günkel, Kehl
- Italy (5):
  - UOC di Pediatria 1, Milan, Milano
  - Servizio di Igiene e Sanita Pubblica, Sassari, Sassari
  - Dipartimento di Scienze della Salute, Genova
  - Azienda Sanitaria Provinciale di Ragusa, Ragusa
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
- Poland (8):
  - oddzial Neuroinfekcji i Neurologii Dzieciecel, Krakowski Szpital Specjalistyczny im.J ana Pawla II, Krakow, Malopolska
  - Wojewodzka Poradnia Szczepien Ochronnych, Krakow, Malopolska
  - Prywatny Gabinet Lekarski dr n med. Jerzy Brzostek, Dębica
  - NZOZ Praktyka Lekarza Rodzinnego lek.med. Agata Slawin, Kiełczów
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap Sp.z o.o., Lublin
  - NZOZ Praktyka Lekarza Rodzinnego Eskulap Sp.z o.o. ul., Lunlin
  - NZLA Michalkowice Jarosz i Partnerzy Spolka Lekarska, Siemianowice Śląskie
  - NZOZ Praktyka Lekarza Rodzinnego Beata Stecka, Wroclaw
- United Kingdom (4):
  - NIHR Wellcome Trust Clinical Research Facility, Southampton, Hampshire
  - University of Bristol, Clinical Research and Imaging Centre, Bristol
  - St. George's University of London**, London
  - Oxford Vaccine Group, University of Oxford, Oxford

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Absalon J, Anderson AS, Eiden JJ, Balmer P, Harris SL, Jones TR, O'Neill RE, Pregaldien JL, Radley D, Maansson R, Ginis J, Srivastava A, Perez JL. MenB-FHbp Vaccine Protects Against Diverse Meningococcal Strains in Adolescents and Young Adults: Post Hoc Analysis of Two Phase 3 Studies. Infect Dis Ther. 2020 Sep;9(3):641-656. doi: 10.1007/s40121-020-00319-0. Epub 2020 Jul 22. PMID 32700260
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472
- [Derived] Ostergaard L, Vesikari T, Absalon J, Beeslaar J, Ward BJ, Senders S, Eiden JJ, Jansen KU, Anderson AS, York LJ, Jones TR, Harris SL, O'Neill R, Radley D, Maansson R, Pregaldien JL, Ginis J, Staerke NB, Perez JL; B1971009 and B1971016 Trial Investigators. A Bivalent Meningococcal B Vaccine in Adolescents and Young Adults. N Engl J Med. 2017 Dec 14;377(24):2349-2362. doi: 10.1056/NEJMoa1614474. PMID 29236639
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1971009&StudyName=A%20trial%20to%20assess%20the%20lot%20consistency%2C%20safety%2C%20tolerability%20and%20immunogenicity%20of%20bivalent%20rLP2086%20vaccine%20when%20given%20to%20healthy%20sub

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 3596 participants were randomized in this study, out of which 3590 participants received vaccination.
Groups:
- Group 1 rLP2086 Lot 1: Lot 1 on a 0-, 2-, 6- month schedule.
- Group 2 rLP2086 Lot 2: Lot 2 on a 0-, 2-, 6- month schedule
- Group 3 rLP2086 Lot 3: Lot 3 on a 0-, 2-, 6- month schedule
- Group 4 HAV/Saline: Hepatitis A virus vaccine (HAV) on a 0- and 6-month schedule and saline at Month 2.
Period: Overall Study
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3 | Group 4 HAV/Saline
Started | 1508 | 598 | 587 | 897
Completed | 1353 | 537 | 521 | 815
Not Completed | 155 | 61 | 66 | 82
Not completed — Other | 7 | 1 | 4 | 4
Not completed — Medication error without associated AE | 1 | 0 | 0 | 1
Not completed — Pregnancy | 3 | 1 | 2 | 1
Not completed — No longer meets eligibility criteria | 11 | 2 | 3 | 5
Not completed — Adverse Event | 11 | 5 | 6 | 3
Not completed — Protocol deviation | 10 | 5 | 6 | 6
Not completed — Withdrawal by Subject | 33 | 14 | 10 | 12
Not completed — No longer willing to participate | 32 | 13 | 12 | 17
Not completed — Lost to Follow-up | 47 | 20 | 23 | 33

BASELINE CHARACTERISTICS:
Population: Safety population included all the participants who received at least 1 dose of the investigational product (rLP2086 or HAV/saline) and had safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3 | Group 4 HAV/Saline | Total
Number analyzed (Participants) | 1508 | 598 | 587 | 897 | 3590
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.9 (2.6) | 14.0 (2.6) | 13.9 (2.6) | 13.9 (2.6) | 13.9 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 737 | 286 | 274 | 443 | 1740
  Male | 771 | 312 | 313 | 454 | 1850

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With >=4 Fold Rise in Serum Bactericidal Assay Using Human Complement (hSBA) for 4 Primary Strains and Composite Response (hSBA >=Lower Limit of Quantification [LLOQ] for All 4 Primary Strains Combined) for Group 1
Description: Groups 2 and 3 were included for the Lot consistency analysis for primary strains only (hSBA geometric mean titer). The immunogenicity of two MnB strains in lots 1,2,3 were required to test for lot consistency. These data are presented separately in the other endpoints. The data for all the strains in Lot 1 (Group 1) is sufficient to describe the immunogenicity expected with the vaccine. The analytical plan was included in the protocol and agreement was reach with EMA and FDA. Here, N signifies participants with valid and determinate hSBA titers for given strain at specified time point.
Time Frame: One month after third bivalent rLP2086 vaccination
Population: Evaluable immunogenicity population: all eligible participants randomized, who received correct investigational product, had pre/post vaccination blood drawn at pre-specified time points, had valid and determinate assay results for proposed analysis, received no prohibited treatment or prohibited vaccines, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 1279
percentage of participants
  Composite hSBA response (N= 1170) | 83.5 [81.3 to 85.6]
  PMB80[A22] (N= 1225) | 83.2 [81.0 to 85.2]
  PMB2001[A56] (N= 1128) | 90.2 [88.4 to 91.9]
  PMB2948[B24] (N= 1235) | 79.8 [77.4 to 82.0]
  PMB2707[B44] (N= 1203) | 85.9 [83.8 to 87.8]

2. Primary Outcome: hSBA Geometric Mean Titers (GMTs) for Each of the 2 Primary Test Strains Measured 1 Month After the Third Vaccination With Bivalent rLP2086 Vaccine
Time Frame: One month after third bivalent rLP2086 vaccination
Population: Evaluable immunogenicity population. Here, N signifies participants with valid and determinate hSBA titers for the given strain.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 1279 | 519 | 493
titer
  PMB80[A22] (N= 1266, 518, 492) | 86.8 [82.29 to 91.50] | 84.3 [77.54 to 91.68] | 85.1 [78.26 to 92.47]
  PMB2948[B24] (N= 1250, 516, 479) | 24.1 [22.70 to 25.48] | 25.3 [23.08 to 27.72] | 25.2 [23.03 to 27.58]
Statistical Analysis 1: Comparison: Group 1 rLP2086 Lot 1 vs Group 2 rLP2086 Lot 2; PMB80 [A22]: The lot consistency criteria was achieved if the 95% CI for all pairwise GMRs between lots are within (0.5, 2), for the strain PMB80; Test type: Superiority or Other; Ratio of GMTs = 1.03, 95% CI 2-sided [0.93 to 1.14]
Statistical Analysis 2: Comparison: Group 1 rLP2086 Lot 1 vs Group 3 rLP2086 Lot 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio of GMTs = 1.02, 95% CI 2-sided [0.92 to 1.13]
Statistical Analysis 3: Comparison: Group 2 rLP2086 Lot 2 vs Group 3 rLP2086 Lot 3; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio of GMTs = 0.99, 95% CI 2-sided [0.88 to 1.12]
Statistical Analysis 4: Comparison: Group 1 rLP2086 Lot 1 vs Group 2 rLP2086 Lot 2; PMB2948 [B24]: The lot consistency criteria was achieved if the 95% CI for all pairwise GMRs between lots are within (0.5, 2), for the strain PMB2948; Test type: Superiority or Other; Ratio of GMTs = 0.95, 95% CI 2-sided [0.85 to 1.06]
Statistical Analysis 5: Comparison: Group 1 rLP2086 Lot 1 vs Group 3 rLP2086 Lot 3; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Ratio of GMTs = 0.95, 95% CI 2-sided [0.86 to 1.06]
Statistical Analysis 6: Comparison: Group 2 rLP2086 Lot 2 vs Group 3 rLP2086 Lot 3; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Ratio of GMTs = 1.00, 95% CI 2-sided [0.88 to 1.14]

3. Primary Outcome: Percentage of Participants Reporting Local Reactions (LRs) Within 7 Days After First Vaccination
Time Frame: Within 7 Days after first vaccination
Population: Safety population for first vaccination included all participants who received the first dose of investigational product (rLP2086 or HAV) and for whom safety information was available from first vaccination until prior to second vaccination. Here,number of participants analyzed signifies participants with known values after the first vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- rLP2086 (Lots 1-3): Commercial lots 1, 2 and 3 on a 0-, 2-, 6-months schedule.
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2681 | 890
percentage of participants
  Pain at injection site: Any | 86.7 [85.4 to 88.0] | 47.0 [43.6 to 50.3]
  Pain at injection site: Mild | 41.1 [39.2 to 43.0] | 36.5 [33.3 to 39.8]
  Pain at injection site: Moderate | 40.7 [38.8 to 42.5] | 9.9 [8.0 to 12.0]
  Pain at injection site: Severe | 5.0 [4.2 to 5.9] | 0.6 [0.2 to 1.3]
  Redness: Any | 16.2 [14.8 to 17.7] | 1.3 [0.7 to 2.3]
  Redness: Mild | 5.6 [4.7 to 6.5] | 1.2 [0.6 to 2.2]
  Redness: Moderate | 8.8 [7.7 to 9.9] | 0.1 [0.0 to 0.6]
  Redness: Severe | 1.9 [1.4 to 2.5] | 0.0 [0.0 to 0.4]
  Swelling: Any | 18.0 [16.5 to 19.5] | 2.2 [1.4 to 3.4]
  Swelling: Mild | 8.5 [7.4 to 9.6] | 1.8 [1.0 to 2.9]
  Swelling: Moderate | 8.8 [7.7 to 9.9] | 0.4 [0.1 to 1.1]
  Swelling: Severe | 0.7 [0.5 to 1.1] | 0.0 [0.0 to 0.4]

4. Primary Outcome: Percentage of Participants Reporting Local Reactions (LRs) Within 7 Days After Second Vaccination
Time Frame: Within 7 Days after second vaccination
Population: Safety population for second vaccination included all participants who received the second dose of investigational product (rLP2086 or saline), for whom safety information was available from second vaccination until prior to third vaccination.Here,number of participants analyzed signifies participants with known values after second vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2545 | 843
percentage of participants
  Pain at injection site: Any | 77.7 [76.0 to 79.3] | 15.2 [12.8 to 17.8]
  Pain at injection site: Mild | 39.4 [37.5 to 41.3] | 12.3 [10.2 to 14.7]
  Pain at injection site: Moderate | 33.2 [31.4 to 35.1] | 2.7 [1.7 to 4.1]
  Pain at injection site: Severe | 5.1 [4.2 to 6.0] | 0.1 [0.0 to 0.7]
  Redness: Any | 12.5 [11.2 to 13.8] | 0.6 [0.2 to 1.4]
  Redness: Mild | 5.2 [4.4 to 6.2] | 0.6 [0.2 to 1.4]
  Redness: Moderate | 6.1 [5.2 to 7.1] | 0.0 [0.0 to 0.4]
  Redness: Severe | 1.1 [0.8 to 1.6] | 0.0 [0.0 to 0.4]
  Swelling: Any | 13.9 [12.5 to 15.3] | 0.6 [0.2 to 1.4]
  Swelling: Mild | 6.3 [5.4 to 7.3] | 0.5 [0.1 to 1.2]
  Swelling: Moderate | 7.3 [6.4 to 8.4] | 0.1 [0.0 to 0.7]
  Swelling: Severe | 0.2 [0.1 to 0.5] | 0.0 [0.0 to 0.4]

5. Primary Outcome: Percentage of Participants Reporting Local Reactions (LRs) Within 7 Days After Third Vaccination
Time Frame: Within 7 Days after third vaccination
Population: Safety population for third vaccination included all participants who received third dose of investigational product (rLP2086 or HAV) and for whom safety information was available from third vaccination until post third-vaccination blood draw.Here,number of participants analyzed signifies participants with known values after third vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2421 | 821
percentage of participants
  Pain at injection site: Any | 76.0 [74.2 to 77.7] | 34.0 [30.7 to 37.3]
  Pain at injection site: Mild | 34.1 [32.2 to 36.0] | 23.8 [20.9 to 26.8]
  Pain at injection site: Moderate | 36.5 [34.6 to 38.5] | 9.9 [7.9 to 12.1]
  Pain at injection site: Severe | 5.4 [4.5 to 6.4] | 0.4 [0.1 to 1.1]
  Redness: Any | 13.9 [12.5 to 15.3] | 1.1 [0.5 to 2.1]
  Redness: Mild | 4.9 [4.1 to 5.8] | 1.0 [0.4 to 1.9]
  Redness: Moderate | 6.8 [5.8 to 7.9] | 0.1 [0.0 to 0.7]
  Redness: Severe | 2.2 [1.6 to 2.9] | 0.0 [0.0 to 0.4]
  Swelling: Any | 15.4 [14.0 to 16.9] | 0.9 [0.3 to 1.7]
  Swelling: Mild | 7.9 [6.8 to 9.0] | 0.7 [0.3 to 1.6]
  Swelling: Moderate | 6.8 [5.8 to 7.9] | 0.1 [0.0 to 0.7]
  Swelling: Severe | 0.7 [0.4 to 1.1] | 0.0 [0.0 to 0.4]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After First Vaccination
Description: Here, N signifies participants with known values reporting specific characteristic.
Time Frame: Within 7 Days after first vaccination
Population: Safety population for first vaccination included all participants who received the first dose of investigational product (rLP2086 or HAV) and for whom safety information was available from first vaccination until prior to second vaccination.Here,number of participants analyzed signifies participants with known values after the first vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2681 | 890
percentage of participants
  Fever >=38 degrees C(N=2679, 890) | 6.4 [5.5 to 7.4] | 1.9 [1.1 to 3.0]
  Fever 38 to <38.5 degreesC(N=2679, 890) | 4.0 [3.3 to 4.8] | 1.3 [0.7 to 2.3]
  Fever 38.5 to<39 degrees C(N=2679, 890) | 1.9 [1.5 to 2.5] | 0.3 [0.1 to 1.0]
  Fever 39 to 40 degrees C(N=2679, 890) | 0.5 [0.3 to 0.8] | 0.2 [0.0 to 0.8]
  Fever >40 degrees C(N=2679, 890) | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.4]
  Vomiting:Any(N=2681,890) | 3.7 [3.0 to 4.5] | 1.9 [1.1 to 3.0]
  Vomiting:Mild(N=2681,890) | 2.8 [2.2 to 3.5] | 1.7 [0.9 to 2.8]
  Vomiting:Moderate(N=2681,890) | 0.9 [0.6 to 1.4] | 0.2 [0.0 to 0.8]
  Vomiting:Severe(N=2681,890) | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.4]
  Diarrhea:Any(N=2681,890) | 10.6 [9.5 to 11.9] | 12.1 [10.1 to 14.5]
  Diarrhea:Mild(N=2681,890) | 9.1 [8.0 to 10.3] | 10.9 [8.9 to 13.1]
  Diarrhea:Moderate(N=2681,890) | 1.3 [0.9 to 1.8] | 1.1 [0.5 to 2.1]
  Diarrhea:Severe(N=2681,890) | 0.3 [0.1 to 0.5] | 0.1 [0.0 to 0.6]
  Headache:Any(N=2681,890) | 51.8 [49.9 to 53.8] | 37.2 [34.0 to 40.5]
  Headache:Mild(N=2681,890) | 28.7 [27.0 to 30.5] | 24.0 [21.3 to 27.0]
  Headache:Moderate(N=2681,890) | 21.0 [19.4 to 22.6] | 12.5 [10.4 to 14.8]
  Headache:Severe(N=2681,890) | 2.2 [1.6 to 2.8] | 0.7 [0.2 to 1.5]
  Fatigue:Any(N=2681,890) | 54.0 [52.1 to 55.9] | 40.3 [37.1 to 43.6]
  Fatigue:Mild(N=2681,890) | 27.8 [26.1 to 29.5] | 23.5 [20.7 to 26.4]
  Fatigue:Moderate(N=2681,890) | 23.2 [21.6 to 24.8] | 15.2 [12.9 to 17.7]
  Fatigue:Severe(N=2681,890) | 3.0 [2.4 to 3.7] | 1.7 [0.9 to 2.8]
  Chills:Any(N=2681,890) | 25.3 [23.7 to 27.0] | 17.2 [14.8 to 19.8]
  Chills:Mild(N=2681,890) | 16.2 [14.8 to 17.6] | 13.3 [11.1 to 15.7]
  Chills:Moderate(N=2681,890) | 8.0 [7.0 to 9.1] | 3.5 [2.4 to 4.9]
  Chills:Severe(N=2681,890) | 1.2 [0.8 to 1.7] | 0.4 [0.1 to 1.1]
  Muscle pain:Any(N=2681,890) | 24.4 [22.8 to 26.1] | 19.2 [16.7 to 22.0]
  Muscle pain:Mild(N=2681,890) | 13.2 [11.9 to 14.5] | 13.5 [11.3 to 15.9]
  Muscle pain:Moderate(N=2681,890) | 10.1 [9.0 to 11.3] | 5.4 [4.0 to 7.1]
  Muscle pain:Severe(N=2681,890) | 1.2 [0.8 to 1.6] | 0.3 [0.1 to 1.0]
  Joint pain:Any(N=2681,890) | 21.9 [20.4 to 23.5] | 13.6 [11.4 to 16.0]
  Joint pain:Mild(N=2681,890) | 11.8 [10.6 to 13.1] | 8.3 [6.6 to 10.3]
  Joint pain:Moderate(N=2681,890) | 8.7 [7.7 to 9.8] | 4.6 [3.3 to 6.2]
  Joint pain:Severe(N=2681,890) | 1.4 [1.0 to 1.9] | 0.7 [0.2 to 1.5]
  Antipyretic medication(N=2681,890) | 20.7 [19.2 to 22.3] | 10.4 [8.5 to 12.6]

7. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After Second Vaccination
Description: Here, N signifies participants with known values reporting specific characteristic.
Time Frame: Within 7 Days after second vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2545 | 843
percentage of participants
  Fever >=38 degrees C(N=2540, 840) | 2.0 [1.5 to 2.6] | 1.5 [0.8 to 2.6]
  Fever 38 to <38.5 degreesC(N=2540, 840) | 1.2 [0.8 to 1.7] | 0.7 [0.3 to 1.5]
  Fever 38.5 to<39 degrees C(N=2540, 840) | 0.7 [0.4 to 1.1] | 0.7 [0.3 to 1.5]
  Fever 39 to 40 degrees C(N=2540, 840) | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.7]
  Fever >40 degrees C(N=2540, 840) | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.4]
  Vomiting:Any(N=2545, 843) | 2.2 [1.6 to 2.8] | 1.4 [0.7 to 2.5]
  Vomiting:Mild(N=2545, 843) | 1.7 [1.3 to 2.3] | 1.1 [0.5 to 2.0]
  Vomiting:Moderate(N=2545, 843) | 0.4 [0.2 to 0.8] | 0.4 [0.1 to 1.0]
  Vomiting:Severe(N=2545, 843) | 0.0 [0.0 to 0.1] | 0.0 [0.0 to 0.4]
  Diarrhea:Any(N=2545, 843) | 7.6 [6.6 to 8.7] | 9.1 [7.3 to 11.3]
  Diarrhea:Mild(N=2545, 843) | 6.2 [5.3 to 7.2] | 7.6 [5.9 to 9.6]
  Diarrhea:Moderate(N=2545, 843) | 1.3 [0.9 to 1.8] | 1.2 [0.6 to 2.2]
  Diarrhea:Severe(N=2545, 843) | 0.1 [0.0 to 0.3] | 0.4 [0.1 to 1.0]
  Headache:Any(N=2545, 843) | 37.8 [35.9 to 39.8] | 28.1 [25.1 to 31.3]
  Headache:Mild(N=2545, 843) | 20.2 [18.7 to 21.8] | 15.7 [13.3 to 18.3]
  Headache:Moderate(N=2545, 843) | 16.0 [14.6 to 17.5] | 10.9 [8.9 to 13.2]
  Headache:Severe(N=2545, 843) | 1.7 [1.2 to 2.2] | 1.5 [0.8 to 2.6]
  Fatigue:Any(N=2545, 843) | 38.3 [36.4 to 40.2] | 26.3 [23.4 to 29.4]
  Fatigue:Mild(N=2545, 843) | 20.6 [19.0 to 22.2] | 13.2 [11.0 to 15.6]
  Fatigue:Moderate(N=2545, 843) | 15.8 [14.4 to 17.3] | 11.7 [9.6 to 14.1]
  Fatigue:Severe(N=2545, 843) | 1.9 [1.4 to 2.5] | 1.4 [0.7 to 2.5]
  Chills:Any(N=2545, 843) | 16.0 [14.6 to 17.4] | 10.3 [8.3 to 12.6]
  Chills:Mild(N=2545, 843) | 10.6 [9.4 to 11.9] | 8.1 [6.3 to 10.1]
  Chills:Moderate(N=2545, 843) | 4.8 [4.0 to 5.7] | 1.8 [1.0 to 2.9]
  Chills:Severe(N=2545, 843) | 0.6 [0.3 to 1.0] | 0.5 [0.1 to 1.2]
  Muscle pain:Any(N=2545, 843) | 17.8 [16.3 to 19.3] | 10.3 [8.3 to 12.6]
  Muscle pain:Mild(N=2545, 843) | 8.7 [7.6 to 9.8] | 5.2 [3.8 to 6.9]
  Muscle pain:Moderate(N=2545, 843) | 7.9 [6.8 to 9.0] | 4.5 [3.2 to 6.1]
  Muscle pain:Severe(N=2545, 843) | 1.2 [0.8 to 1.7] | 0.6 [0.2 to 1.4]
  Joint pain:Any(N=2545, 843) | 16.7 [15.3 to 18.2] | 9.1 [7.3 to 11.3]
  Joint pain:Mild(N=2545, 843) | 8.4 [7.4 to 9.6] | 5.0 [3.6 to 6.7]
  Joint pain:Moderate(N=2545, 843) | 7.5 [6.5 to 8.6] | 3.4 [2.3 to 4.9]
  Joint pain:Severe(N=2545, 843) | 0.8 [0.5 to 1.2] | 0.7 [0.3 to 1.5]
  Antipyretic medication(N=2545, 843) | 13.6 [12.3 to 15.0] | 8.9 [7.1 to 11.0]

8. Primary Outcome: Percentage of Participants Reporting Systemic Events (SEs) and Antipyretic Use Within 7 Days After Third Vaccination
Description: Here, N signifies participants with known values reporting specific characteristic.
Time Frame: Within 7 Days after third vaccination
Population: Safety population for third vaccination included all participants who received third dose of investigational product (rLP2086 or HAV) and for whom safety information was available from third vaccination until post third-vaccination blood draw. Here, number of participants analyzed signifies participants with known values after third vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2421 | 821
percentage of participants
  Fever >=38 degrees C(N=2414, 819) | 2.7 [2.1 to 3.4] | 2.3 [1.4 to 3.6]
  Fever 38 to <38.5degreesC(N=2414, 819) | 1.8 [1.3 to 2.4] | 1.3 [0.7 to 2.4]
  Fever 38.5 to<39 degrees C(N=2414, 819) | 0.6 [0.3 to 1.0] | 0.4 [0.1 to 1.1]
  Fever 39 to 40 degrees C(N=2414, 819) | 0.3 [0.1 to 0.6] | 0.5 [0.1 to 1.2]
  Fever >40 degrees C(N=2414, 819) | 0.0 [0.0 to 0.2] | 0.1 [0.0 to 0.7]
  Vomiting:Any(N=2421, 821) | 1.7 [1.3 to 2.3] | 2.2 [1.3 to 3.4]
  Vomiting:Mild(N=2421, 821) | 1.4 [1.0 to 2.0] | 1.7 [0.9 to 2.8]
  Vomiting:Moderate(N=2421, 821) | 0.3 [0.1 to 0.6] | 0.5 [0.1 to 1.2]
  Vomiting:Severe(N=2421, 821) | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.4]
  Diarrhea:Any(N=2421, 821) | 7.7 [6.7 to 8.9] | 7.6 [5.8 to 9.6]
  Diarrhea:Mild(N=2421, 821) | 6.4 [5.5 to 7.5] | 6.2 [4.7 to 8.1]
  Diarrhea:Moderate(N=2421, 821) | 1.0 [0.6 to 1.5] | 1.1 [0.5 to 2.1]
  Diarrhea:Severe(N=2421, 821) | 0.3 [0.1 to 0.6] | 0.2 [0.0 to 0.9]
  Headache:Any(N=2421, 821) | 35.4 [33.5 to 37.4] | 24.8 [21.9 to 28.0]
  Headache:Mild(N=2421, 821) | 18.9 [17.3 to 20.5] | 13.5 [11.3 to 16.1]
  Headache:Moderate(N=2421, 821) | 15.2 [13.8 to 16.7] | 10.4 [8.4 to 12.6]
  Headache:Severe(N=2421, 821) | 1.3 [0.9 to 1.9] | 1.0 [0.4 to 1.9]
  Fatigue:Any(N=2421, 821) | 35.9 [34.0 to 37.9] | 24.4 [21.5 to 27.4]
  Fatigue:Mild(N=2421, 821) | 18.4 [16.9 to 20.0] | 13.5 [11.3 to 16.1]
  Fatigue:Moderate(N=2421, 821) | 15.2 [13.8 to 16.7] | 10.0 [8.0 to 12.2]
  Fatigue:Severe(N=2421, 821) | 2.3 [1.8 to 3.0] | 0.9 [0.3 to 1.7]
  Chills:Any(N=2421, 821) | 13.1 [11.7 to 14.5] | 8.3 [6.5 to 10.4]
  Chills:Mild(N=2421, 821) | 8.7 [7.6 to 9.9] | 6.5 [4.9 to 8.4]
  Chills:Moderate(N=2421, 821) | 3.8 [3.1 to 4.7] | 1.7 [0.9 to 2.8]
  Chills:Severe(N=2421, 821) | 0.5 [0.3 to 0.9] | 0.1 [0.0 to 0.7]
  Muscle pain:Any(N=2421, 821) | 17.6 [16.1 to 19.1] | 11.1 [9.0 to 13.4]
  Muscle pain:Mild(N=2421, 821) | 9.5 [8.4 to 10.8] | 6.6 [5.0 to 8.5]
  Muscle pain:Moderate(N=2421, 821) | 7.2 [6.2 to 8.3] | 4.3 [3.0 to 5.9]
  Muscle pain:Severe(N=2421, 821) | 0.8 [0.5 to 1.3] | 0.2 [0.0 to 0.9]
  Joint pain:Any(N=2421, 821) | 16.0 [14.6 to 17.5] | 8.9 [7.0 to 11.1]
  Joint pain:Mild(N=2421, 821) | 8.9 [7.8 to 10.1] | 5.5 [4.0 to 7.3]
  Joint pain:Moderate(N=2421, 821) | 5.9 [5.0 to 6.9] | 3.0 [2.0 to 4.5]
  Joint pain:Severe(N=2421, 821) | 1.2 [0.8 to 1.8] | 0.4 [0.1 to 1.1]
  Antipyretic medication(N=2421, 821) | 12.7 [11.4 to 14.1] | 6.8 [5.2 to 8.8]

9. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: Safety population for first vaccination included all participants who received the first dose of investigational product (rLP2086 or HAV) and for whom safety information was available from first vaccination until prior to second vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.26 [0.1 to 0.5] | 0.33 [0.1 to 1.0]

10. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: Safety population for second vaccination included all participants who received the second dose of investigational product (rLP2086 or saline) and for whom safety information was available from second vaccination until prior to third vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2570 | 860
percentage of participants | 0.23 [0.1 to 0.5] | 0.23 [0.0 to 0.8]

11. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: Safety population for third vaccination included all participants who received the third dose of investigational product (rLP2086 or HAV) and for whom safety information was available from third vaccination until post third-vaccination blood draw.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2462 | 835
percentage of participants | 0.32 [0.1 to 0.6] | 0.36 [0.1 to 1.0]

12. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.78 [0.5 to 1.2] | 0.89 [0.4 to 1.7]

13. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 1.49 [1.1 to 2.0] | 1.90 [1.1 to 3.0]

14. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) During the Follow-Up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: Safety population: all participants who had at least 1 dose investigational product (rLP2086 or HAV/saline) for whom safety information was available from after post third-vaccination blood draw to 6 months after last study vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2524 | 839
percentage of participants | 0.44 [0.2 to 0.8] | 0.60 [0.2 to 1.4]

15. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE) Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 1.89 [1.4 to 2.5] | 2.45 [1.5 to 3.7]

16. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 5.27 [4.5 to 6.2] | 6.69 [5.1 to 8.5]

17. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2570 | 860
percentage of participants | 5.91 [5.0 to 6.9] | 6.51 [5.0 to 8.4]

18. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2462 | 835
percentage of participants | 5.81 [4.9 to 6.8] | 7.43 [5.7 to 9.4]

19. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Within 30 Days After Any Vaccination
Time Frame: Within 30 days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 14.18 [12.9 to 15.6] | 16.61 [14.2 to 19.2]

20. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 25.29 [23.7 to 27.0] | 27.87 [25.0 to 30.9]

21. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE During the Follow-Up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or HAV/saline) for whom safety information was available from after post-vaccination 3 blood draw to 6 months after last study vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2524 | 839
percentage of participants | 15.61 [14.2 to 17.1] | 16.92 [14.4 to 19.6]

22. Primary Outcome: Percentage of Participants With at Least 1 Medically Attended AE Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 32.38 [30.6 to 34.2] | 35.56 [32.4 to 38.8]

23. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.00 [0.0 to 0.1] | 0.11 [0.0 to 0.6]

24. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Second Vaccination
Time Frame: 30 days after second vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2570 | 860
percentage of participants | 0.08 [0.0 to 0.3] | 0.12 [0.0 to 0.6]

25. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2462 | 835
percentage of participants | 0.12 [0.0 to 0.4] | 0.00 [0.0 to 0.4]

26. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Within 30 Days After Any Vaccination
Time Frame: Within 30 Days After any Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.19 [0.1 to 0.4] | 0.22 [0.0 to 0.8]

27. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.37 [0.2 to 0.7] | 0.56 [0.2 to 1.3]

28. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition During the Follow-Up Phase
Time Frame: From 1 month after third vaccination up to 6 months after the third vaccination
Population: Safety population: all participants who had at least 1 dose of investigational product (rLP2086 or HAV/saline) for whom safety information was available from after post third-vaccination blood draw to 6 months after last study vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2524 | 839
percentage of participants | 0.20 [0.1 to 0.5] | 0.60 [0.2 to 1.4]

29. Primary Outcome: Percentage of Participants With at Least 1 Newly Diagnosed Chronic Medical Condition Throughout the Study Period
Time Frame: From the first vaccination up to 6 month after the third vaccination
Population: Safety population included all participants who received at least 1 dose of the investigational product and had safety information available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.56 [0.3 to 0.9] | 1.11 [0.5 to 2.0]

30. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) WIthin 30 Days After First Vaccination
Time Frame: Within 30 days after first vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 9.51 [8.4 to 10.7] | 10.70 [8.8 to 12.9]

31. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Second Vaccination
Time Frame: Within 30 days after second vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2570 | 860
percentage of participants | 11.48 [10.3 to 12.8] | 12.67 [10.5 to 15.1]

32. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Within 30 Days After Third Vaccination
Time Frame: Within 30 days after third vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2462 | 835
percentage of participants | 9.91 [8.8 to 11.2] | 10.78 [8.8 to 13.1]

33. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event Within 30 Days After Any Vaccination
Time Frame: Within 30 Days after any vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 25.32 [23.7 to 27.0] | 26.76 [23.9 to 29.8]

34. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 40.74 [38.9 to 42.6] | 43.70 [40.4 to 47.0]

35. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After First Vaccination
Time Frame: Within 30 minutes after first vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2693 | 897
percentage of participants | 0.1 [0.0 to 0.4] | 0.2 [0.0 to 0.8]

36. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Second Vaccination
Time Frame: Within 30 minutes after second vaccination
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2570 | 860
percentage of participants | 0.2 [0.0 to 0.4] | 0.1 [0.0 to 0.6]

37. Primary Outcome: Percentage of Participants Reporting at Least 1 Immediate AE After Third Vaccination
Time Frame: Within 30 minutes after third vaccination
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 2462 | 835
percentage of participants | 0.1 [0.0 to 0.3] | 0.0 [0.0 to 0.4]

38. Primary Outcome: Number of Days Participant's Missed School or Work Due to AE During the Vaccination Phase
Time Frame: From the first vaccination up to 1 month after the third vaccination
Population: Safety population included all the participants who received at least 1 dose of the investigational product (rLP2086 or HAV/saline) and had safety data available. Here, number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | rLP2086 (Lots 1-3) | Group 4 HAV/Saline
Number analyzed (Participants) | 539 | 195
days | 3.9 (6.56) | 4.0 (5.19)

39. Secondary Outcome: Percentage of Participants With hSBA Titers >=LLOQ for 10 Secondary Strains Before First Vaccination and 1 Month After Third Bivalent rLP2086 Vaccination for Group 1
Description: Groups 2 and 3 were included for the Lot consistency analysis for primary strains only (hSBA geometric mean titer). The immunogenicity of two MnB strains in lots 1, 2, 3 were required to test for lot consistency. These data are presented separately in the other endpoints. The data for all the strains in Lot 1 (Group 1) is sufficient to describe the immunogenicity expected with the vaccine. The analytical plan was included in the protocol and agreement was reach with EMA and FDA.
Time Frame: Before first vaccination, 1 month after third vaccination
Population: Evaluable immunogenicity population. Here, number of participants analyzed signifies participants with valid and determinate hSBA titers for the given strain. Here, N signifies participants with valid and determinate hSBA titers for the given strain at the specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 300
percentage of participants
  PMB3175[A29]:Before Vaccination 1 (N= 269) | 17.5 [13.1 to 22.5]
  PMB3175[A29]:1 Month after Vaccination 3 (N= 278) | 98.6 [96.4 to 99.6]
  PMB3010[A06]:Before Vaccination 1 (N= 277) | 9.4 [6.2 to 13.5]
  PMB3010[A06]:1 Month after Vaccination 3 (N= 280) | 95.7 [92.6 to 97.8]
  PMB3040[A07]:Before Vaccination 1 (N= 269) | 43.1 [37.1 to 49.3]
  PMB3040[A07]:1 Month after Vaccination 3 (N= 280) | 96.4 [93.5 to 98.3]
  PMB824[A12]: Before Vaccination 1 (N= 280) | 3.9 [2.0 to 6.9]
  PMB824[A12]:1 Month after Vaccination 3 (N= 277) | 75.1 [69.6 to 80.1]
  PMB1672[A15]:Before Vaccination 1 (N= 270) | 20.7 [16.1 to 26.1]
  PMB1672[A15]:1 Month after Vaccination 3 (N= 266) | 87.2 [82.6 to 91.0]
  PMB1989[A19]:Before Vaccination 1 (N= 274) | 11.3 [7.8 to 15.7]
  PMB1989[A19]:1 Month after Vaccination 3 (N= 275) | 92.7 [89.0 to 95.5]
  PMB1256[B03]:Before Vaccination 1 (N= 280) | 4.3 [2.2 to 7.4]
  PMB1256[B03]:1 Month after Vaccination 3 (N= 279) | 92.5 [88.7 to 95.3]
  PMB866[B09]:Before Vaccination 1 (N= 277) | 15.2 [11.2 to 19.9]
  PMB866[B09]:1 Month after Vaccination 3 (N= 276) | 86.2 [81.6 to 90.1]
  PMB431[B15]:Before Vaccination 1 (N= 275) | 28.7 [23.5 to 34.5]
  PMB431[B15]:1 Month after Vaccination 3 (N= 281) | 98.2 [95.9 to 99.4]
  PMB648[B16]:Before Vaccination 1 (N= 276) | 7.6 [4.8 to 11.4]
  PMB648[B16]:1 Month after Vaccination 3 (N= 278) | 81.7 [76.6 to 86.0]

40. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, >=1:128 for Each of the 10 Secondary Strains, Before Vaccination 1 and 1 Month After the Third Bivalent rLP2086 Vaccination for Group 1
Description: as for outcome 39
Time Frame: Before first vaccination, 1 month after third vaccination (Vac)
Population: as for outcome 39
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 300
percentage of participants
  Before Vaccination 1: PMB3175[A29] 1:4 (N=269) | 19.0 [14.5 to 24.2]
  1 month after Vac 3: PMB3175[A29] 1:4 (N=278) | 98.6 [96.4 to 99.6]
  Before Vaccination 1: PMB3175[A29] 1:8 (N=269) | 17.5 [13.1 to 22.5]
  1 month after Vac 3: PMB3175[A29] 1:8 (N=278) | 98.6 [96.4 to 99.6]
  Before Vaccination 1: PMB3175[A29] 1:16 (N=269) | 16.7 [12.5 to 21.7]
  1 month after Vac 3: PMB3175[A29] 1:16 (N=278) | 98.6 [96.4 to 99.6]
  Before Vaccination 1: PMB3175[A29] 1:32 (N=269) | 10.8 [7.3 to 15.1]
  1 month after Vac 3: PMB3175[A29] 1:32 (N=278) | 97.5 [94.9 to 99.0]
  Before Vaccination 1: PMB3175[A29] 1:64 (N=269) | 4.8 [2.6 to 8.1]
  1 month after Vac 3: PMB3175[A29] 1:64 (N=278) | 86.0 [81.3 to 89.8]
  Before Vaccination 1: PMB3175[A29] 1:128 (N=269) | 1.1 [0.2 to 3.2]
  1 month after Vac 3: PMB3175[A29] 1:128 (N=278) | 52.2 [46.1 to 58.2]
  Before Vaccination 1: PMB3010[A06] 1:4 (N=277) | 9.7 [6.5 to 13.9]
  1 month after Vac 3: PMB3010[A06] 1:4 (N=280) | 96.1 [93.1 to 98.0]
  Before Vaccination 1: PMB3010[A06] 1:8 (N=277) | 9.7 [6.5 to 13.9]
  1 month after Vac 3: PMB3010[A06] 1:8 (N=280) | 96.1 [93.1 to 98.0]
  Before Vaccination 1: PMB3010[A06] 1:16 (N=277) | 9.4 [6.2 to 13.5]
  1 month after Vac 3: PMB3010[A06] 1:16 (N=280) | 95.7 [92.6 to 97.8]
  Before Vaccination 1: PMB3010[A06] 1:32 (N=277) | 6.1 [3.6 to 9.6]
  1 month after Vac 3: PMB3010 [A06] 1:32 (N=280) | 93.6 [90.0 to 96.1]
  Before Vaccination 1: PMB3010[A06] 1:64 (N=277) | 2.9 [1.3 to 5.6]
  1 month after Vac 3: PMB3010[A06] 1:64 (N=280) | 78.2 [72.9 to 82.9]
  Before Vaccination 1: PMB3010[A06] 1:128 (N=277) | 1.4 [0.4 to 3.7]
  1 month after Vac 3: PMB3010[A06] 1:128 (N=280) | 44.3 [38.4 to 50.3]
  Before Vaccination 1: PMB3040[A07] 1:4 (N=269) | 43.1 [37.1 to 49.3]
  1 month after Vac 3: PMB3040[A07] 1:4 (N=280) | 96.4 [93.5 to 98.3]
  Before Vaccination 1: PMB3040[A07] 1:8 (N=269) | 43.1 [37.1 to 49.3]
  1 month after Vac 3: PMB3040[A07] 1:8 (N=280) | 96.4 [93.5 to 98.3]
  Before Vaccination 1: PMB3040[A07] 1:16 (N=269) | 42.8 [36.8 to 48.9]
  1 month after Vac 3: PMB3040[A07] 1:16 (N=280) | 96.4 [93.5 to 98.3]
  Before Vaccination 1: PMB3040[A07] 1:32 (N=269) | 37.2 [31.4 to 43.3]
  1 month after Vac 3: PMB3040[A07] 1:32 (N=280) | 93.6 [90.0 to 96.1]
  Before Vaccination 1: PMB3040[A07] 1:64 (N=269) | 21.6 [16.8 to 27.0]
  1 month after Vac 3: PMB3040[A07] 1:64 (N=280) | 78.2 [72.9 to 82.9]
  Before Vaccination 1: PMB3040[A07] 1:128 (N=269) | 5.6 [3.2 to 9.0]
  1 month after Vac 3: PMB3040[A07] 1:128 (N=280) | 30.4 [25.0 to 36.1]
  Before Vaccination 1: PMB824[A12] 1:4 (N=280) | 5.4 [3.0 to 8.7]
  1 month after Vac 3: PMB824[A12] 1:4 (N=277) | 77.6 [72.2 to 82.4]
  Before Vaccination 1: PMB824[A12] 1:8 (N=280) | 4.6 [2.5 to 7.8]
  1 month after Vac 3: PMB824[A12] 1:8 (N=277) | 77.3 [71.9 to 82.1]
  Before Vaccination 1: PMB824[A12] 1:16 (N=280) | 3.9 [2.0 to 6.9]
  1 month after Vac 3: PMB824[A12] 1:16 (N=277) | 75.1 [69.6 to 80.1]
  Before Vaccination 1: PMB824[A12] 1:32 (N=280) | 2.5 [1.0 to 5.1]
  1 month after Vac 3: PMB824[A12] 1:32 (N=277) | 51.3 [45.2 to 57.3]
  Before Vaccination 1: PMB824[A12] 1:64 (N=280) | 0.0 [0.0 to 1.3]
  1 month after Vac 3: PMB824[A12] 1:64 (N=277) | 19.5 [15.0 to 24.7]
  Before Vaccination 1: PMB824[A12] 1:128 (N=280) | 0.0 [0.0 to 1.3]
  1 month after Vac 3: PMB824[A12] 1:128 (N=277) | 1.8 [0.6 to 4.2]
  Before Vaccination 1: PMB1672[A15] 1:4 (N=270) | 22.6 [17.7 to 28.1]
  1 month after Vac 3: PMB1672[A15] 1:4 (N=266) | 87.2 [82.6 to 91.0]
  Before Vaccination 1: PMB1672[A15] 1:8 (N=270) | 20.7 [16.1 to 26.1]
  1 month after Vac 3: PMB1672[A15] 1:8 (N=266) | 87.2 [82.6 to 91.0]
  Before Vaccination 1: PMB1672[A15] 1:16 (N=270) | 17.0 [12.8 to 22.1]
  1 month after Vac 3: PMB1672[A15] 1:16 (N=266) | 85.0 [80.1 to 89.0]
  Before Vaccination 1: PMB1672[A15] 1:32 (N=270) | 13.3 [9.5 to 18.0]
  1 month after Vac 3: PMB1672[A15] 1:32 (N=266) | 71.4 [65.6 to 76.8]
  Before Vaccination 1: PMB1672[A15] 1:64 (N=270) | 3.7 [1.8 to 6.7]
  1 month after Vac 3: PMB1672[A15] 1:64 (N=266) | 40.2 [34.3 to 46.4]
  Before Vaccination 1: PMB1672[A15] 1:128 (N=270) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB1672[A15] 1:128 (N=266) | 10.5 [7.1 to 14.9]
  Before Vaccination 1: PMB1989[A19] 1:4 (N=274) | 20.8 [16.2 to 26.1]
  1 month after Vac 3: PMB1989[A19] 1:4 (N=275) | 93.8 [90.3 to 96.4]
  Before Vaccination 1: PMB1989[A19] 1:8 (N=274) | 18.6 [14.2 to 23.7]
  1 month after Vac 3: PMB1989[A19] 1:8 (N=275) | 93.8 [90.3 to 96.4]
  Before Vaccination 1: PMB1989[A19] 1:16 (N=274) | 11.3 [7.8 to 15.7]
  1 month after Vac 3: PMB1989[A19] 1:16 (N=275) | 92.7 [89.0 to 95.5]
  Before Vaccination 1: PMB1989[A19] 1:32 (N=274) | 5.8 [3.4 to 9.3]
  1 month after Vac 3: PMB1989[A19] 1:32 (N=275) | 85.5 [80.7 to 89.4]
  Before Vaccination 1: PMB1989[A19] 1:64 (N=274) | 1.8 [0.6 to 4.2]
  1 month after Vac 3: PMB1989[A19] 1:64 (N=275) | 60.0 [53.9 to 65.8]
  Before Vaccination 1: PMB1989[A19] 1:128 (N=274) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB1989[A19] 1:128 (N=275) | 33.1 [27.6 to 39.0]
  Before Vaccination 1: PMB1256[B03] 1:4 (N=280) | 5.0 [2.8 to 8.2]
  1 month after Vac 3: PMB1256[B03] 1:4 (N=279) | 92.5 [88.7 to 95.3]
  Before Vaccination 1: PMB1256[B03] 1:8 (N=280) | 4.3 [2.2 to 7.4]
  1 month after Vac 3: PMB1256[B03] 1:8 (N=279) | 92.5 [88.7 to 95.3]
  Before Vaccination 1: PMB1256[B03] 1:16 (N=280) | 4.3 [2.2 to 7.4]
  1 month after Vac 3: PMB1256[B03] 1:16 (N=279) | 92.1 [88.3 to 95.0]
  Before Vaccination 1: PMB1256[B03] 1:32 (N=280) | 3.9 [2.0 to 6.9]
  1 month after Vac 3: PMB1256[B03] 1:32 (N=279) | 81.4 [76.3 to 85.8]
  Before Vaccination 1: PMB1256[B03] 1:64 (N=280) | 2.9 [1.2 to 5.6]
  1 month after Vac 3: PMB1256[B03] 1:64 (N=279) | 60.6 [54.6 to 66.3]
  Before Vaccination 1: PMB1256[B03] 1:128 (N=280) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB1256[B03] 1:128 (N=279) | 29.4 [24.1 to 35.1]
  Before Vaccination 1: PMB866[B09] 1:4 (N=277) | 15.5 [11.5 to 20.3]
  1 month after Vac 3: PMB866[B09] 1:4 (N=276) | 86.6 [82.0 to 90.4]
  Before Vaccination 1: PMB866[B09] 1:8 (N=277) | 15.2 [11.2 to 19.9]
  1 month after Vac 3: PMB866[B09] 1:8 (N=276) | 86.2 [81.6 to 90.1]
  Before Vaccination 1: PMB866[B09] 1:16 (N=277) | 13.7 [9.9 to 18.3]
  1 month after Vac 3: PMB866[B09] 1:16 (N=276) | 83.7 [78.8 to 87.9]
  Before Vaccination 1: PMB866[B09] 1:32 (N=277) | 8.7 [5.6 to 12.6]
  1 month after Vac 3: PMB866[B09] 1:32 (N=276) | 54.0 [47.9 to 60.0]
  Before Vaccination 1: PMB866[B09] 1:64 (N=277) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB866[B09] 1:64 (N=276) | 21.4 [16.7 to 26.7]
  Before Vaccination 1: PMB866[B09] 1:128 (N=277) | 0.0 [0.0 to 1.3]
  1 month after Vac 3: PMB866[B09] 1:128 (N=276) | 4.3 [2.3 to 7.5]
  Before Vaccination 1: PMB431[B15] 1:4 (N=275) | 30.5 [25.2 to 36.4]
  1 month after Vac 3: PMB431[B15] 1:4 (N=281) | 98.2 [95.9 to 99.4]
  Before Vaccination 1: PMB431[B15] 1:8 (N=275) | 28.7 [23.5 to 34.5]
  1 month after Vac 3: PMB431[B15] 1:8 (N=281) | 98.2 [95.9 to 99.4]
  Before Vaccination 1: PMB431[B15] 1:16 (N=275) | 27.6 [22.4 to 33.3]
  1 month after Vac 3: PMB431[B15] 1:16 (N=281) | 97.5 [94.9 to 99.0]
  Before Vaccination 1: PMB431[B15] 1:32 (N=275) | 21.8 [17.1 to 27.2]
  1 month after Vac 3: PMB431[B15] 1:32 (N=281) | 85.1 [80.3 to 89.0]
  Before Vaccination 1: PMB431[B15] 1:64 (N=275) | 8.4 [5.4 to 12.3]
  1 month after Vac 3: PMB431[B15] 1:64 (N=281) | 56.2 [50.2 to 62.1]
  Before Vaccination 1: PMB431[B15] 1:128 (N=275) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB431[B15] 1:128 (N=281) | 19.2 [14.8 to 24.3]
  Before Vaccination 1: PMB648[B16] 1:4 (N=276) | 8.7 [5.7 to 12.7]
  1 month after Vac 3: PMB648[B16] 1:4 (N=278) | 82.7 [77.8 to 87.0]
  Before Vaccination 1: PMB648[B16] 1:8 (N=276) | 7.6 [4.8 to 11.4]
  1 month after Vac 3: PMB648[B16] 1:8 (N=278) | 81.7 [76.6 to 86.0]
  Before Vaccination 1: PMB648[B16] 1:16 (N=276) | 7.6 [4.8 to 11.4]
  1 month after Vac 3: PMB648[B16] 1:16 (N=278) | 79.9 [74.7 to 84.4]
  Before Vaccination 1: PMB648[B16] 1:32 (N=276) | 6.2 [3.6 to 9.7]
  1 month after Vac 3: PMB648[B16] 1:32 (N=278) | 54.0 [47.9 to 59.9]
  Before Vaccination 1: PMB648[B16] 1:64 (N=276) | 1.8 [0.6 to 4.2]
  1 month after Vac 3: PMB648[B16] 1:64 (N=278) | 24.1 [19.2 to 29.6]
  Before Vaccination 1: PMB648[B16] 1:128 (N=276) | 0.4 [0.0 to 2.0]
  1 month after Vac 3: PMB648[B16] 1:128 (N=278) | 5.8 [3.3 to 9.2]

41. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) for Each of the 10 Secondary Strains Before First Vaccination and 1 Month After the Third Bivalent rLP2086 Vaccination for Group 1
Description: as for outcome 39
Time Frame: Before first vaccination, 1 month after third vaccination
Population: Evaluable immunogenicity population. Here, number of participants analyzed signifies participants with valid and determinate hSBA titers for the given strain. Here, N signifies participants with valid and determinate assay results for the given antigen or strain.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 300
titer
  PMB3175[A29]:Before Vaccination 1 (N= 269) | 5.7 [5.16 to 6.28]
  PMB3175[A29]:1 Month after Vaccination 3 (N= 278) | 93.5 [84.79 to 103.09]
  PMB3010[A06]:Before Vaccination 1 (N= 277) | 9.3 [8.68 to 9.91]
  PMB3010[A06]:1 Month after Vaccination 3 (N= 280) | 78.6 [70.94 to 87.08]
  PMB3040[A07]:Before Vaccination 1 (N= 269) | 11.4 [9.75 to 13.23]
  PMB3040[A07]:1 Month after Vaccination 3 (N= 280) | 63.5 [57.93 to 69.66]
  PMB824[A12]: Before Vaccination 1 (N= 280) | 8.4 [8.14 to 8.59]
  PMB824[A12]:1 Month after Vaccination 3 (N= 277) | 22.3 [20.37 to 24.45]
  PMB1672[A15]:Before Vaccination 1 (N= 270) | 5.9 [5.32 to 6.46]
  PMB1672[A15]:1 Month after Vaccination 3 (N= 266) | 31.0 [27.43 to 35.07]
  PMB1989[A19]:Before Vaccination 1 (N= 274) | 9.1 [8.70 to 9.62]
  PMB1989[A19]:1 Month after Vaccination 3 (N= 275) | 57.6 [51.30 to 64.60]
  PMB1256[B03]:Before Vaccination 1 (N= 280) | 4.5 [4.19 to 4.75]
  PMB1256[B03]:1 Month after Vaccination 3 (N= 279) | 51.7 [45.36 to 58.89]
  PMB866[B09]:Before Vaccination 1 (N= 277) | 5.2 [4.82 to 5.62]
  PMB866[B09]:1 Month after Vaccination 3 (N= 276) | 22.9 [20.48 to 25.63]
  PMB431[B15]:Before Vaccination 1 (N= 275) | 7.3 [6.49 to 8.23]
  PMB431[B15]:1 Month after Vaccination 3 (N= 281) | 47.7 [43.66 to 52.16]
  PMB648[B16]:Before Vaccination 1 (N= 276) | 4.7 [4.39 to 5.05]
  PMB648[B16]:1 Month after Vaccination 3 (N= 278) | 22.1 [19.60 to 24.98]

42. Secondary Outcome: Percentage of Participants Achieving Composite hSBA Titer >=Lower Limit of Quantitation for All 4 Primary Strains Before First Vaccination and 1 Month After Second Bivalent rLP2086 Vaccination for Group 1
Description: Groups 2 and 3 were included for the Lot consistency analysis for primary strains only (hSBA geometric mean titer). The immunogenicity of two MnB strains in lots 1, 2 ,3 were required to test for lot consistency. These data are presented separately in the other endpoints. The data for all the strains in Lot 1 (Group 1) is sufficient to describe the immunogenicity expected with the vaccine. The analytical plan was included in the protocol and agreement was reach with EMA and FDA.
Time Frame: Before vaccination 1, 1 Month after Vaccination 2
Population: Evaluable immunogenicity population. Here, N signifies participants valid and determinate hSBA results on all 4 strains at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 1279
percentage of participants
  Before First Vaccination (N= 1088) | 1.1 [0.6 to 1.9]
  1 Month after Vaccination 2 (N= 1122) | 54.1 [51.1 to 57.0]

43. Secondary Outcome: Percentage of Participants Achieving at Least a 4-Fold Increase in hSBA Titer for Each of the 4 Primary Strains Before First Vaccination to 1 Month After the Second Bivalent rLP2086 Vaccination for Group 1
Description: as for outcome 39
Time Frame: One month after second Bivalent rLP2086 vaccination
Population: Evaluable immunogenicity population. Here, N signifies participants with valid and determinate hSBA titers for the given strain at both the specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1
Number analyzed (Participants) | 1279
percentage of participants
  PMB80[A22] (N=1223) | 73.8 [71.2 to 76.2]
  PMB2001[A56] (N=1122) | 84.8 [82.5 to 86.8]
  PMB2948[B24] (N=1201) | 56.2 [53.3 to 59.0]
  PMB2707[B44] (N=1197) | 55.9 [53.0 to 58.7]

44. Secondary Outcome: Percentage of Participants Achieving at Least a 4-Fold Increase in hSBA Titer for 2 Primary Strains Before First Vaccination to 1 Month After the Second and Third Bivalent rLP2086 Vaccination
Time Frame: One month after second, third vaccination
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 519 | 493
percentage of participants
  PMB80[A22]:1Month after Vaccination 2 (N=493, 473) | 71.2 [67.0 to 75.2] | 74.6 [70.5 to 78.5]
  PMB80[A22]:1Month after Vaccination 3 (N=501, 478) | 83.8 [80.3 to 86.9] | 86.0 [82.5 to 89.0]
  PMB2948[B24]:1Month after Vaccination 2(N=490,463) | 56.7 [52.2 to 61.2] | 56.8 [52.2 to 61.4]
  PMB2948[B24]:1Month after Vaccination 3(N=507,472) | 76.5 [72.6 to 80.2] | 78.4 [74.4 to 82.0]

45. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) for 4 Primary Test Strains and for 2 Primary Test Strains and Before First Vaccination and 1 Month After the Second Bivalent rLP2086 Vaccination
Time Frame: Before vaccination (Vac) 1, 1 Month after Vac 2
Population: Evaluable immunogenicity population. Here, N signifies participants with valid and determinate hSBA titers for the given strain at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 1279 | 519 | 493
titer
  PMB80[A22]: Before Vac 1 (N=1238, 502, 479) | 12.6 [12.08 to 13.14] | 12.9 [12.06 to 13.79] | 12.2 [11.43 to 13.04]
  PMB80[A22]: 1 Month after Vac 2 (N=1263, 510, 487) | 50.4 [47.76 to 53.09] | 47.7 [43.82 to 51.97] | 49.6 [45.58 to 53.99]
  PMB2001[A56]: Before Vac 1 (N=1135, 0, 0) | 8.4 [7.80 to 9.05] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  PMB2001[A56]: 1 Month after Vac 2 (N=1222, 0, 0) | 131.2 [124.03 to 138.70] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  PMB2948[B24]: Before Vac 1 (N=1264, 510, 486) | 4.5 [4.37 to 4.60] | 4.6 [4.43 to 4.85] | 4.6 [4.43 to 4.88]
  PMB2948[B24]: 1 Month after Vac 2 (N=1216,499,470) | 14.3 [13.45 to 15.31] | 14.5 [13.23 to 15.98] | 15.2 [13.75 to 16.85]
  PMB2707[B44]: Before Vac 1 (N=1230, 0, 0) | 4.3 [4.17 to 4.34] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  PMB2707[B44]: 1 Month after Vac 2 (N=1204, 0, 0) | 17.1 [15.80 to 18.60] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.

46. Secondary Outcome: Percentage of Participants With hSBA Titers >=LLOQ for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination
Time Frame: Before Vaccination (Vac) 1, 1 Month after Vac 2, 3
Population: Evaluable immunogenicity population. Here N signifies participants with valid and determinate hSBA titers for the given strain at the specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 1279 | 519 | 493
percentage of participants
  Before Vac 1: PMB80[A22] 1:16(N=1238, 502, 479) | 33.2 [30.6 to 35.9] | 34.9 [30.7 to 39.2] | 31.7 [27.6 to 36.1]
  1 month afterVac2:PMB80[A22]1:16(N=1263,510,487) | 94.3 [92.9 to 95.5] | 92.7 [90.1 to 94.8] | 94.7 [92.3 to 96.5]
  1 month after Vac3:PMB80[A22]1:16(N=1266, 518,492) | 97.8 [96.8 to 98.5] | 97.3 [95.5 to 98.5] | 98.2 [96.6 to 99.2]
  Before Vac 1: PMB2001[A56] 1:8(N=1135, 0, 0) | 27.5 [24.9 to 30.2] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3 | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3
  1 month after Vac2:PMB2001[A56]1:8(N=1222, 0, 0) | 99.1 [98.4 to 99.5] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3 | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3
  1 month after Vac3:PMB2001[A56]1:8(N=1229, 0, 0) | 99.5 [98.9 to 99.8] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3 | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3
  Before Vac 1: PMB2948[B24]1:8(N=1264, 510, 486) | 6.4 [5.1 to 7.9] | 8.6 [6.3 to 11.4] | 8.4 [6.1 to 11.3]
  1 monthafterVac2:PMB2948[B24]1:8(N=1216,499,470) | 66.4 [63.6 to 69.0] | 70.1 [65.9 to 74.1] | 70.2 [65.9 to 74.3]
  1 monthafterVac3:PMB2948[B24]1:8(N=1250,516,479) | 87.1 [85.1 to 88.9] | 87.6 [84.4 to 90.3] | 90.0 [86.9 to 92.5]
  Before Vac 1: PMB2707[B44] 1:8(N=1230, 0, 0) | 3.6 [2.6 to 4.8] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:8(N=1204, 0, 0) | 64.0 [61.3 to 66.8] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2707[B44]1:8(N=1210, 0, 0) | 89.3 [87.4 to 90.9] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.

47. Secondary Outcome: Percentage of Participants With hSBA Titers >=1:4,>=1:8,>=1:16,>=1:32,>=1:64,>=1:128 for Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination
Description: Results for PMB80[A22] 1:16, PMB2001[A56] 1:8, PMB2948[B24] 1:8 and PMB2707[B44] 1:8 are reported under secondary outcome measure 'Percentage of Participants With hSBA Titers >=LLOQ for 4 Primary Test Strains Before First Vaccination, 1 Month After Second and Third Bivalent rLP2086 Vaccination.
Time Frame: Before Vaccination (Vac) 1, 1 Month after Vac 2, 3
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 1279 | 519 | 493
percentage of participants
  Before Vac 1:PMB80[A22] 1:4(N=1238, 502, 479) | 36.2 [33.5 to 38.9] | 39.6 [35.3 to 44.1] | 36.7 [32.4 to 41.2]
  1 month after Vac2:PMB80[A22]1:4(N=1263, 510, 487) | 94.9 [93.6 to 96.1] | 93.7 [91.3 to 95.7] | 95.5 [93.2 to 97.1]
  1 month after Vac3:PMB80[A22]1:4(N=1266, 518, 492) | 97.9 [97.0 to 98.7] | 98.1 [96.5 to 99.1] | 98.4 [96.8 to 99.3]
  Before Vac 1: PMB80[A22] 1:8(N=1238, 502, 479) | 34.8 [32.2 to 37.5] | 39.0 [34.8 to 43.5] | 34.7 [30.4 to 39.1]
  1 month after Vac2:PMB80[A22]1:8(N=1263, 510, 487) | 94.7 [93.3 to 95.9] | 93.5 [91.0 to 95.5] | 95.5 [93.2 to 97.1]
  1 month after Vac3:PMB80[A22]1:8(N=1266, 518, 492) | 97.9 [97.0 to 98.7] | 98.1 [96.5 to 99.1] | 98.4 [96.8 to 99.3]
  Before Vac 1: PMB80[A22] 1:32(N=1238, 502, 479) | 20.9 [18.7 to 23.3] | 21.7 [18.2 to 25.6] | 19.8 [16.4 to 23.7]
  1 month after Vac2:PMB80[A22]1:32(N=1263, 510,487) | 81.9 [79.7 to 84.0] | 79.4 [75.6 to 82.8] | 80.7 [76.9 to 84.1]
  1 month after Vac3:PMB80[A22]1:32(N=1266,518,492) | 93.0 [91.4 to 94.3] | 92.1 [89.4 to 94.3] | 93.1 [90.5 to 95.2]
  Before Vac 1: PMB80[A22] 1:64(N=1238, 502, 479) | 8.5 [7.0 to 10.2] | 9.6 [7.1 to 12.5] | 5.4 [3.6 to 7.9]
  1 month after Vac2:PMB80[A22]1:64(N=1263,510,487) | 51.8 [49.0 to 54.6] | 49.6 [45.2 to 54.0] | 51.5 [47.0 to 56.1]
  1 month after Vac3:PMB80[A22]1:64(N=1266,518,492) | 75.3 [72.8 to 77.6] | 75.5 [71.5 to 79.1] | 73.6 [69.4 to 77.4]
  Before Vac 1: PMB80[A22] 1:128(N=1238, 502,479) | 2.0 [1.3 to 3.0] | 2.0 [1.0 to 3.6] | 2.5 [1.3 to 4.3]
  1 month after Vac2:PMB80[A22]1:128(N=1263,510,487) | 24.5 [22.1 to 26.9] | 23.5 [19.9 to 27.5] | 24.4 [20.7 to 28.5]
  1 month after Vac3:PMB80[A22]1:128(N=1266,518,492) | 48.3 [45.6 to 51.1] | 46.3 [42.0 to 50.7] | 49.2 [44.7 to 53.7]
  Before Vac 1: PMB2001[A56] 1:4(N=1135, 0, 0) | 29.5 [26.9 to 32.3] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2001[A56]1:4(N=1222, 0, 0) | 99.1 [98.4 to 99.5] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2001[A56]1:4(N=1229, 0, 0) | 99.5 [98.9 to 99.8] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2001[A56] 1:16(N=1135, 0, 0) | 27.4 [24.8 to 30.1] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2001[A56]1:16(N=1222,0,0) | 99.1 [98.4 to 99.5] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2001[A56]1:16(N=1229,0,0) | 99.4 [98.8 to 99.8] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2001[A56] ] 1:32(N=1135, 0, 0) | 25.6 [23.0 to 28.2] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2001[A56] 1:32(N=1222,0,0) | 97.2 [96.1 to 98.1] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2001[A56]1:32(N=1229,0,0) | 98.6 [97.8 to 99.2] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2001[A56] 1:64(N=1135, 0, 0) | 17.1 [14.9 to 19.4] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month afterVac2:PMB2001[A56]1:64(N=1222,0,0) | 89.4 [87.6 to 91.1] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2001[A56]1:64(N=1229,0,0) | 94.5 [93.0 to 95.7] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2001[A56] 1:128(N=1135, 0, 0) | 6.4 [5.1 to 8.0] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2001[A56]1:128(N=1222,0,0) | 63.4 [60.6 to 66.1] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  1 month afterVac3:PMB2001[A56]1:128(N=1229,0,0) | 82.9 [80.7 to 85.0] | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001 [A56] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2948[B24] 1:4(N=1264, 510, 486) | 6.8 [5.5 to 8.3] | 10.2 [7.7 to 13.2] | 9.5 [7.0 to 12.4]
  1 month after Vac2:PMB2948[B24]1:4(N=1216,499,470) | 69.2 [66.6 to 71.8] | 72.9 [68.8 to 76.8] | 74.0 [69.8 to 78.0]
  1 month after Vac3:PMB2948[B24]1:4(N=1250,516,479) | 88.9 [87.0 to 90.6] | 89.9 [87.0 to 92.4] | 91.6 [88.8 to 94.0]
  Before Vac 1: PMB2948[B24] 1:16(N=1264, 510, 486) | 5.4 [4.2 to 6.8] | 7.5 [5.3 to 10.1] | 7.0 [4.9 to 9.6]
  1 month afterVac2:PMB2948[B24]1:16(N=1216,499,470) | 60.0 [57.2 to 62.8] | 61.5 [57.1 to 65.8] | 62.1 [57.6 to 66.5]
  1 month afterVac3:PMB2948[B24]1:16(N=1250,516,479) | 82.6 [80.4 to 84.7] | 81.2 [77.6 to 84.5] | 83.1 [79.4 to 86.3]
  Before Vac 1: PMB2948[B24] 1:32(N=1264, 510, 486) | 2.8 [2.0 to 3.9] | 3.9 [2.4 to 6.0] | 3.7 [2.2 to 5.8]
  1 month afterVac2:PMB2948[B24]1:32(N=1216,499,470) | 33.0 [30.3 to 35.7] | 34.5 [30.3 to 38.8] | 35.5 [31.2 to 40.0]
  1 month afterVac3:PMB2948[B24]1:32(N=1250,516,479) | 52.1 [49.3 to 54.9] | 54.8 [50.4 to 59.2] | 54.1 [49.5 to 58.6]
  Before Vac 1:PMB2948[B24] 1:64(N=1264, 510, 486) | 1.3 [0.7 to 2.0] | 1.2 [0.4 to 2.5] | 1.9 [0.9 to 3.5]
  1 monthafterVac2:PMB2948[B24]1:64(N=1216,499,470) | 15.3 [13.3 to 17.4] | 13.0 [10.2 to 16.3] | 15.3 [12.2 to 18.9]
  1 month afterVac3:PMB2948[B24]1:64(N=1250,516,479) | 22.8 [20.5 to 25.2] | 27.5 [23.7 to 31.6] | 25.3 [21.4 to 29.4]
  Before Vac 1:PMB2948[B24] 1:128(N=1264, 510,486) | 0.5 [0.2 to 1.0] | 0.2 [0.0 to 1.1] | 0.4 [0.0 to 1.5]
  1 monthafterVac2:PMB2948[B24]1:128(N=1216,499,470) | 6.2 [4.9 to 7.7] | 5.2 [3.4 to 7.5] | 7.0 [4.9 to 9.7]
  1 monthafterVac3:PMB2948[B24]1:128(N=1250,516,479) | 8.9 [7.4 to 10.6] | 11.2 [8.6 to 14.3] | 8.6 [6.2 to 11.4]
  Before Vac 1: PMB2707[B44] 1:4(N=1230, 0, 0) | 4.6 [3.5 to 5.9] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:4(N=1204, 0,0) | 66.7 [64.0 to 69.4] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2707[B44]1:4(N=1210, 0,0) | 90.4 [88.6 to 92.0] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2707[B44] 1:16(N=1230, 0, 0) | 3.0 [2.1 to 4.1] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:16(N=1204,0,0) | 57.7 [54.9 to 60.5] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month afterVac3:PMB2707[B44]1:16(N=1210,0, 0) | 86.8 [84.7 to 88.6] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1: PMB2707[B44] 1:32(N=1230, 0, 0) | 1.6 [1.0 to 2.5] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:32(N=1204,0,0) | 39.0 [36.3 to 41.9] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2707[B44]1:32(N=1210,0,0) | 71.6 [68.9 to 74.1] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1:PMB2707[B44] 1:64(N=1230, 0, 0) | 0.7 [0.3 to 1.3] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:64(N=1204,0,0) | 23.3 [21.0 to 25.8] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2707[B44]1:64(N=1210,0,0) | 54.5 [51.7 to 57.4] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  Before Vac 1:PMB2707[B44] 1:128(N=1230, 0, 0) | 0.2 [0.0 to 0.6] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac2:PMB2707[B44]1:128(N=1204,0,0) | 13.0 [11.2 to 15.1] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.
  1 month after Vac3:PMB2707[B44]1:128(N=1210,0,0) | 35.0 [32.4 to 37.8] | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707 [B44] was not planned to be analyzed for Group 2 and Group 3.

48. Secondary Outcome: Percentage of Participants Achieving at Least a 3-Fold Increase in hSBA Titer for 4 Primary Test Strains and for Primary Test Starins Before First Vaccination to 1 Month After Third Bivalent rLP2086 Vaccination
Time Frame: One month after third bivalent rLP2086 vaccination
Population: Data was not reported because 3-fold rise analyses was not performed as per change in planned analysis.
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 0 | 0 | 0

49. Secondary Outcome: Percentage of Participants Achieving at Least a 2-Fold Increase in hSBA Titer for 4 Primary Test Strains and for 2 Primary Test Starins Before First Vaccination to 1 Month After the Third Bivalent rLP2086 Vaccination
Time Frame: One month after third bivalent rLP2086 vaccination (Vac)
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3
Number analyzed (Participants) | 1279 | 519 | 493
percentage of participants
  PMB80[A22]: 1 Month after Vac 3(N=1225, 501, 478) | 91.43 [89.7 to 92.9] | 92.02 [89.3 to 94.2] | 93.51 [90.9 to 95.6]
  PMB2001[A56]: 1 Month after Vac 3(N=1128, 0, 0) | 95.04 [93.6 to 96.2] | NA [NA to NA] — PMB2001[A56] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2001[A56] was not planned to be analyzed for Group 2 and Group 3.
  PMB2948[B24]: 1 Month after Vac 3(N=1235, 507,472) | 81.05 [78.8 to 83.2] | 79.09 [75.3 to 82.6] | 80.93 [77.1 to 84.4]
  PMB2707[B44]: 1 Month after Vac 3(N=1203, 0, 0) | 86.62 [84.6 to 88.5] | NA [NA to NA] — PMB2707[B44] was not planned to be analyzed for Group 2 and Group 3. | NA [NA to NA] — PMB2707[B44] was not planned to be analyzed for Group 2 and Group 3.

ADVERSE EVENTS:
Time Frame: AEs/SAEs: recorded from first vaccination through 6 months after third vaccination. Participants recorded pre-specified reactogenicity events (local reactions, systemic events) in electronic diary within 7 days after first, second and third vaccination
Description: All AEs collected on case report form are shown below as having been collected via non-systematic assessment. All events reported via electronic diary (reactogenicity events) are shown below as having been collected via systematic assessment. Reactogenicity events are grouped by all severities and doses combined.
Arm/Group | Group 1 rLP2086 Lot 1 | Group 2 rLP2086 Lot 2 | Group 3 rLP2086 Lot 3 | Group 4 HAV/Saline
Serious Adverse Events (participants affected / at risk) | 22/1508 | 10/598 | 19/587 | 22/897
Other Adverse Events (participants affected / at risk) | 1410/1508 | 547/598 | 542/587 | 655/897
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 rLP2086 Lot 1 (N=1508) | Group 2 rLP2086 Lot 2 (N=598) | Group 3 rLP2086 Lot 3 (N=587) | Group 4 HAV/Saline (N=897)
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 4
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 2
Anorexia nervosa (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Borderline personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Group 1 rLP2086 Lot 1 (N=1508) | Group 2 rLP2086 Lot 2 (N=598) | Group 3 rLP2086 Lot 3 (N=587) | Group 4 HAV/Saline (N=897)
Abdominal pain (Gastrointestinal disorders) | 29 | 5 | 9 | 8
Diarrhea (Gastrointestinal disorders) | 15 | 6 | 3 | 15
Vomiting (Gastrointestinal disorders) | 14 | 4 | 2 | 12
Nausea (Gastrointestinal disorders) | 10 | 7 | 3 | 7
Pyrexia (General disorders) | 18 | 8 | 5 | 8
Fatigue (General disorders) | 5 | 3 | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 105 | 53 | 45 | 70
Pharyngitis (Infections and infestations) | 69 | 21 | 24 | 43
Nasopharyngitis (Infections and infestations) | 59 | 32 | 32 | 32
Gastroenteritis (Infections and infestations) | 43 | 25 | 19 | 25
Sinusitis (Infections and infestations) | 34 | 19 | 14 | 22
Bronchitis (Infections and infestations) | 27 | 6 | 10 | 19
Otitis media (Infections and infestations) | 19 | 11 | 11 | 16
Pharyngitis streptococcal (Infections and infestations) | 21 | 6 | 10 | 13
Influenza (Infections and infestations) | 19 | 9 | 8 | 9
Acute sinusitis (Infections and infestations) | 18 | 8 | 7 | 7
Urinary tract infection (Infections and infestations) | 18 | 5 | 10 | 7
Viral infection (Infections and infestations) | 15 | 8 | 4 | 12
Viral pharyngitis (Infections and infestations) | 19 | 4 | 2 | 9
Tonsillitis (Infections and infestations) | 10 | 7 | 3 | 10
Otitis externa (Infections and infestations) | 8 | 9 | 3 | 9
Otitis media acute (Infections and infestations) | 8 | 6 | 2 | 10
Gastroenteritis viral (Infections and infestations) | 8 | 3 | 1 | 9
Fall (Injury, poisoning and procedural complications) | 42 | 19 | 9 | 20
Ligament sprain (Injury, poisoning and procedural complications) | 36 | 14 | 8 | 24
Contusion (Injury, poisoning and procedural complications) | 20 | 7 | 6 | 19
Muscle strain (Injury, poisoning and procedural complications) | 7 | 5 | 1 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 11 | 3 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 3 | 2 | 12
Headache (Nervous system disorders) | 42 | 21 | 15 | 23
Dizziness (Nervous system disorders) | 5 | 6 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 9 | 7 | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 7 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 3 | 5 | 6
Acne (Skin and subcutaneous tissue disorders) | 14 | 6 | 14 | 11
Dermatitis contact (Skin and subcutaneous tissue disorders) | 14 | 7 | 5 | 5
Pain at injection site -Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 1403/1504 | 544/597 | 541/585 | 525
Redness -Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 365/1504 | 136/597 | 145/585 | 21/893
Swelling -Any (reactogenicity event) (Skin and subcutaneous tissue disorders) | 416/1504 | 161/597 | 158/585 | 26/893
Fever >=38.0 degrees C -Any (reactogenicity event) (General disorders) | 154/1504 | 52/597 | 57/585 | 46/892
Vomiting -Any (reactogenicity event) (General disorders) | 110/1504 | 31/597 | 44/585 | 41/893
Diarrhea-Any (reactogenicity event) (General disorders) | 294/1504 | 114/597 | 117/585 | 187/893
Headache -Any (reactogenicity event) (General disorders) | 1032/1504 | 379/597 | 392/585 | 477/893
Fatigue -Any (reactogenicity event) (General disorders) | 1011/1504 | 380/597 | 369/585 | 454/893
Chills-Any (reactogenicity event) (General disorders) | 566/1504 | 183/597 | 225/585 | 227/893
Muscle pain -Any (reactogenicity event) (General disorders) | 598/1504 | 205/597 | 210/585 | 254/893
Joint pain -Any (reactogenicity event) (General disorders) | 532/1504 | 170/597 | 191/585 | 209/893

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.